CLINICAL TRIAL: NCT04078945
Title: Risk Factors of Shoulder Injuries in Youth Volleyball Players : Prospective Study
Brief Title: Risk Factors of Shoulder Injuries in Youth Volleyball Players
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Physiotherapist, University of Liege
Other Study IDs: Risk factors volleyball
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Shoulder Injuries
Keywords: strength; risk factors; youth volleyball players
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Shoulder injuries are usual in volleyball players. Nowadays, few prospective studies assessed risk factors of shoulder injuries in this sport. So, the objective of this study is to assess the risk factors of injuries in youth volleyball players. For that purpose, the following factors will be taken into consideration : shoulder internal/external rotators strength, shoulder range of motion, scapular dyskinesis, functional tests (medicine ball throw and upper quarter Y balance test), training load and psychosocial factors (POMS questionnaire).

DETAILED DESCRIPTION:
About 100 youth volleyball players (13-20 years), playing at least 8 hours volleyball in a week will be included in the study.

At the beginning of the 2019-2020 season, they will have to take part at the following evaluations :

1. Clinical evaluation :

   * Scapular dyskinesis assessment (normal, subtle abnormality and obvious abnormality)
   * Scapular upward rotation at 0°, 45°,90° and 120° with an inclinometer.
   * Rounded shoulder posture
   * Posterior shoulder stiffness
   * Internal/external rotation range of motion (at 90° of abduction)
2. Medicine ball throw :

   From a cocking position, players have to throw a 800g medicine ball as far as possible (3 trials). Only the best result will be retained for analysis. Volunteers have 2 minutes of rest between trials.
3. Upper Quarter Y Balance Test :

   In a facial drop position, the purpose of this test is to bring the plastic board as far as possible in the 3 directions (supero-lateral, infero-lateral, medial). 3 trials are performed by each subject and only the best test is kept for analysis. A rest period of one minute is provided between tests to avoid fatigue.
4. Strength assessment (isokinetic test) :

   Internal and external rotators strength (concentric 60°/s, eccentric 60°/s and concentric 240°/s) are measured with an isokinetic device (Cybex Norm) at 90° of abduction.
5. Psychosocial factors assessment :

Players will have to fill in POMS questionnaire (65 questions), that give information about stress and well-being.

After that, players will be followed during all the 2019-2020 season and will have to fill in a form each month about the potential injuries they had during the previous month.

ELIGIBILITY:
Inclusion Criteria:

* age between 13 and 20
* to play volleyball at least 8 hours in a week

Exclusion Criteria:

There are no exclusion criteria

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Youth volleyball players, playing at good level in Wallonia (Belgium) will be included in the study
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Shoulder internal/external rotation range of motion | 1 month
  Range of motion will be measured in degrees
Scapular dyskinesis | 1 month
  "yes/no" method
Internal/external rotators strength | 1 month
  Strength of internal and external rotators will be assessed in concentric (60°/s and 240°/s) and in eccentric (60°/s) modes with an isokinetic device (Cybex Norm).
Upper Quarter Y Balance test | 1 month
  The score obtained will be measured in cm and normalized by upperlimb length
Medicine ball throw | 1 month
  A 800g medicine throw will have to be thrown as far as possible and the score will be measured in meters
Psychosocial factors | up to 8 months
  Questionnaire POMS will have to be filled in by the participants each month
Shoulder injuries | up to 8 months
  Participants will have to mention each month the injuries or pain they had during the previous month at shoulder location

CONTACTS AND LOCATIONS:
Overall Officials: Camille Tooth, Principal Investigator — University of Liege
Locations (1):
- Belgium, Wallonia, Liège, Belgium